CLINICAL TRIAL: NCT03598192
Title: The Effect and Safety of the Four Points Transversus Abdominis Plane Block Under the Ultrasound Guidance in Postoperative Analgesia to the Hepatectomy
Brief Title: The Effect and Safety of the Four Points Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Principal Investigator, BINH HUYNH, Department of Anesthesiology, Gia Dinh People Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-2018/CN-HĐĐĐ
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Liver Diseases; Adult Disease
Keywords: Hepatectomy; Transversus abdominis plane block (TAP block); Paravertebral block; Postoperative analgesia; Liver resection
MeSH Terms: conditions — Liver Diseases; Disease | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Intervention Model Description: The TAP group will be performed the four points TAP block under the ultrasound guidance with the ultrasound machine of Logiq E, and linear 12S probe. The participants will be performed TAP block at subcostal and lateral abdominal wall at right and left side with stimuplex needle (sized 18G, length 100 mm). The investigators will approach position between aponeurosis internal oblique and transversus abdominal muscle with in-plane real-time ultrasound technique. The investigators will inject 10 ml of ropivacaine 0.375% at each one. Then, the investigators will access one catheter at TAP at right side to continuously infuse ropivacaine 0.375% during 48 hours after surgery.
  PVB group: the investigators will access one catheter into the right thoracic paravertebral space at T7 before beginning general anesthesia. At the end of surgery, the investigators will inject 20 ml of ropivacaine 0.5% through catheter, and continuously infuse ropivacaine 0.25% during 48 hours after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP group (Experimental): The TAP block is performed under the ultrasound guidance at four points: at subcostal and lateral abdominal wall at right-side and left-side.
  Drug: ropivacaine 0.375% 40 ml (maximum dose <= 3 mg/kg). Maintenance: ropivacaine 0.375% 8 ml/hour during 48 hours.
  Interventions: Procedure: TAP; Drug: Ropivacaine; Drug: Sufentanil
- PVB group (Experimental): The paravertebral block is performed under the ultrasound guidance at T7. Drug: ropivacaine 0.5% 20 ml (maximum dose <= 3 mg/kg). Maintenance: ropivacaine 0.25% 8 ml/hour during 48 hours.
  Interventions: Procedure: PVB; Drug: Ropivacaine; Drug: Sufentanil

INTERVENTIONS:
Procedure: TAP — The TAP group will be performed at four points at abdominis plane with ropivacaine 0.375%
  Other Names: The four points TAP block
  Arms: TAP group
Procedure: PVB — The PVB group will be performed at paravertebral space T7 with ropivacaine 0.5%
  Other Names: The paravertebral block
  Arms: PVB group
Drug: Ropivacaine — Ropivacaine has been treated the both group
  Other Names: have not been specified
Drug: Sufentanil — Sufentanil has been included in Arm/Group Descriptions
  Other Names: Sufentanil PCA

SUMMARY:
The anterior abdominal wall from below the xiphoid to infraumbilical area is dominated by the sensory nerves which originate from the anterior rami of the thoracolumbar spinal nerves from T6-L1. The branches nerves from T7-T12 are between aponeurosis internal oblique and transversus abdominal muscle. They can be approached with the ultrasound guidance at subcostal and lateral abdominal wall position.

The bilateral transversus abdominis plane (TAP) block has been demonstrated effectiveness and safety in postoperative analgesia to the under abdominal surgery. However, the effect of one to the upper abdominal surgery is unclear.

The four points TAP block has been described the first in 2010. The effect of the four points TAP block in postoperative analgesia to the upper abdominal surgery has been reported in recent years. Besides, the effect of thoracic paravertebral block (PVB) in postoperative analgesia to liver resection was also reported. The both techniques have been performing in some studies. The effect and safety of the both techniques have been reported. However, the evidence level is still weak. The investigators need to find a technique, which has effectiveness as well as safety to replace the epidural analgesia, which was confirmed that had many complications, in postoperative analgesia to the hepatectomy.

The investigators hypothesized that the four points TAP block under the ultrasound guidance has more effectiveness than the thoracic paravertebral block in postoperative analgesia to the hepatectomy.

DETAILED DESCRIPTION:
This is a randomized, controlled, no blind, clinical trial. The study was approved by Board of Scientists and Ethic Council in Gia Dinh People Hospital on May 28, 2018. The written informed consent will be obtained from all subjects participating in the trial. The trial will be registered prior to patient enrollment at Gia Dinh People Hospital.

The investigators will select 60 participants who are selective hepatectomy with the "J-shape" incision, II-III of Anesthesiologists Society America (ASA), from 18-75 age. The cases have chronic pain, tolerance opioids, psychology disorder, and allergy opioids or ropivacaine will excluded. All of participants will be randomly divided two groups. There are TAP group and PVB group. Each one has 30 cases.

General anesthesia:

All of cases will be examined, prepared, supplied the study's information on the day before surgical date. The cases, who have enough selective standard, will be selected.

In the operating room, the participants will be performed general anesthesia The participants will be started anesthesia with 1 mg of midazolam, 0.3 mcg/kg of sufentanil, 1-1.5 mg/kg of propofol, and 0.6 mg/kg of rocuronium. Then, the participants will be maintained anesthesia with sevoflurane, sufentanil, and rocuronium. The end of surgery, they will be prevented postoperative nausea and vomiting with 4 mg of ondansetron; and reversed residual of muscle relaxant with sugammadex.

Approaching the transversus abdominal plane:

The technique will be performed at the end of surgery. The TAP group will be performed the four points TAP block under the ultrasound guidance with the ultrasound machine of Logiq E, and linear 12S probe. The participants will be performed TAP block at subcostal and lateral abdominal wall at right and left side with stimuplex needle (sized 18G, length 100 mm). The investigators will approach position between aponeurosis internal oblique and transversus abdominal muscle with in-plane real-time ultrasound technique. The investigators will inject 10 ml of ropivacaine 0.375% at each one. Then, the investigators will access one catheter at TAP at right side to continuously infuse ropivacaine 0.375% during 48 hours after surgery.

Approaching the thoracic paravertebral space:

The investigators will access one catheter into the right thoracic paravertebral space at T7 before beginning general anesthesia. At the end of surgery, we will inject 20 ml of ropivacaine 0.5% through catheter, and continuously infuse ropivacaine 0.25% during 48 hours after surgery.

Patients-controlled analgesia (PCA):

All of participants will be treated postoperative analgesia with sufentanil during 48 hours after operating. The sufentanil will be injected 2 mcg to patients before awaking. Then, the participants will be intravenously infused with PCA (2 mcg of single dosage, 6 minutes of lockout time, and 8 mcg/hour of limited dosage).

The both groups will be intravenously injected 0.2 mg/kg of ketamine at the pre-incisional and post-incisional. After operating, they will be taken 325 mg of paracetamol plus 37.5 mg of tramadol (ultracet tablet) every 8 hours.

Outcomes:

The primary outcome is the consumption of sufentanil (mcg) during 24 hours after operating. The secondary outcomes are the complications of technique, systemic toxicity of ropivacaine, side-effect of sufentanil, and satisfaction of participants.

The complications of the four points TAP block include hematoma in abdominal wall, and puncturing peritoneum. The complications of the thoracic paravertebral block include pneumothorax, and injecting vascular. The hematoma in abdominal wall, puncturing peritoneum, injecting vascular will be observed and recorded by one other anesthesiologist who has not attend the study. The pneumothorax will be diagnosed with the ultrasound by one doctor who is educated the general ultrasound. The systemic toxicity of ropivacaine include central nervous system (CNS) toxicity and cardiovascular toxicity. The signs and symptoms of CNS toxicity include tinnitus, disorientation, and ultimately, seizures. The signs and symptoms of cardiovascular toxicity include hypotension, dysrhythmias, and cardiac arrest. The complications will be treated depending on severity follow the protocol when they occured. The side-effect of sufentanil include sedation, dyspnea, pruritus, and nausea and vomiting. The sedation will be evaluated follow Ramsay scale. The dyspnea is decreasing oxygen saturation by pulse oximetry (SpO2) <= 92%, frequence <= 8 breaths/minute. The satisfaction will be measured follow visual analogue scale (VAS). The VAS scale has from 0 to 10, equivalent to the zero is complete dissatisfaction and the ten is highly satisfaction.

Data processing:

The investigators will process data with SPSS 25.0 (Reg No: 1975-01566-C). The consumption of sufentanil and satisfaction variables will be described by mean (SD) if it is standard distribution, or by median (CI 95%) if it isn't standard distribution. The variables of both groups will be compared by the independent T test or Mann-Whitney test. The quantitive variables will be described by frequency (percentage rate). The investigators will be compared by Chi-square test or exact's Fisher test. The sample size is calculated with 90% of power, and 20% of difference of the consumption of sufentanil of both groups, and 10% of cases losing. The alpha error is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects has selective hepatectomy
* Subjects has had II-III of Anesthesiologists Society Americans

Exclusion Criteria:

* History of chronic pain
* History of tolerance opioids
* History of psychology disorder
* Allergic to ropivacaine or opioids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
The consumption of sulfentanil (mean) | 24 hours
  The consumption of sufentanil is total dose of sufentanil which the participant used during 24 hours. Sufentanil is intravenously infused with PCA, with single dose 1 mcg, limit dose 8 mcg per a hour, and lockout time 5 minutes.

SECONDARY OUTCOMES:
The complications of technique (frequency) | 24 hours
  included injected vascular, hematoma abdominal, pneumothorax, punctured peritoneum, systemic toxicity of ropivacaine
Side-effect of sulfentanil (frequency) | 48 hours
  include sedation, pruritus, nausea and vomiting, dyspnea
Satisfaction (mean) | 24 hours
  evaluated with Visual analogue scale (VAS). VAS is from 0 to 10 that means the minimum satisfaction is 0 score and the maximum satisfaction is 10 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Binh V Huynh, Mr, Study Chair — Nhan dan Gia Dinh Hospital
Locations (1):
- Binh Huynh, Ho Chi Minh City, Ho Chi Minh, Vietnam